CLINICAL TRIAL: NCT05835284
Title: Clinical Data Collection On Advanced CT System
Status: Recruiting | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 199254403; CIV-23-01-042048 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: CT Photon Counting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single Arm: Enrolled subjects will receive a non-diagnostic CT scan on the pre-market, investigational Edge-on Silicon Photon Counting CT device.
  Interventions: Device: Investigational Edge-on Silicon Photon Counting CT device

INTERVENTIONS:
Device: Investigational Edge-on Silicon Photon Counting CT device — Administration of IV contrast material, if applicable, shall be done according to the hospital's SOC. Administration of oral contrast material, if applicable, shall also be done according to the hospital's SOC. Images will then be compared with the previously acquired CT conducted as standard of care. The investigational scan will take approximately 60-120 minutes.

SUMMARY:
The purpose of the study is to evaluate the investigational Edge-on Silicon Photon Counting CT device in a clinical setting.

DETAILED DESCRIPTION:
Images from prior standard of care diagnostic CT exams for these subjects will also be collected. Data collected in this study will be used for technology development, scientific evaluation, marketing and education, and regulatory submissions for future products. This is a pre-market, prospective, open-label, non-randomized, single arm data collection clinical study conducted at one site in Sweden.

ELIGIBILITY:
Inclusion Criteria:

1. 25 years of age or older;
2. Able to sign and date the informed consent form; AND
3. Have undergone a clinically indicated CT exam of the head, neck, chest, abdomen, pelvis, or extremities where images are available within 90 days of investigational scanning.

Exclusion Criteria:

1. Pregnant or lactating;
2. Previously enrolled in this study;
3. For contrast-enhanced CT exams, anyone with known or suspected allergy to iodinated contrast agents;
4. For contrast-enhanced CT exams, anyone with known or suspected renal insufficiency as determined by site medical personnel;
5. Need urgent or emergent care;
6. Have any conditions that, in the opinion of the PI or designee, would interfere with the evaluation of the results or constitute a health hazard for the subject; OR
7. Are unwilling to have GEHC personnel present for the CT exam.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will consist of adults that are 25-years of age or older, and who have undergone prior clinically indicated CT examinations within the past 90 days of at least one of the following anatomical area(s): head, neck, heart, chest, abdomen, pelvis, and extremities. Images from prior standard of care diagnostic CT examinations of these subjects will also be collected.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Data Collection | 12 months
  Raw investigational CT scan data along with standard of care raw CT scan data/images

SECONDARY OUTCOMES:
Safety Information | 12 months
  Type and number of AEs and SAEs
Image Quality | 12 months
  Images created from the raw investigational CT scan data will be scored for image quality using a Likert Scale (1 - Non-Diagnostic to 5 - Excellent Image Quality)

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Thomsen, Study Director — GE Healthcare
Locations (1):
- Karolinska University Hospital, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No